CLINICAL TRIAL: NCT03968497
Title: Impact of Investigator Gender on Perceived Pain Intensity After Acute or Scheduled Surgery
Brief Title: Impact of Gender on Perceived Postoperative Pain
Acronym: G-PAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Gender and pain
Record Dates: First submitted 2019-05-24; First posted 2019-05-30 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Postoperative Pain
Keywords: pain; gender; visual analog scale; numeric rating scale
MeSH Terms: conditions — Pain, Postoperative; Pain; Coitus

STUDY DESIGN:
Intervention Model Description: Half of the patients were first evaluated by the female and then by the male investigator, and the other half the other way around, according to a cross-over study design but with a single group of subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Postoperative pain assessment (Other): Postoperative pain evaluation by a female and a male investigator, respectively at approximately 15-minute intervals.
  Interventions: Other: Postoperative pain assessment with female investigator; Other: Postoperative pain assessment with male investigator

INTERVENTIONS:
Other: Postoperative pain assessment with female investigator — Postoperative pain evaluation by a female investigator by using visual analogue scale, numeric rating scale and Painmatcher®.
  Other Names: Visual analogue scale; Numeric rating scale; Painmatcher®
Other: Postoperative pain assessment with male investigator — Postoperative pain evaluation by a male investigator by using visual analogue scale, numeric rating scale and Painmatcher®.
  Other Names: Visual analogue scale; Numeric rating scale; Painmatcher®

SUMMARY:
Postoperative pain is a common problem after surgical procedures with many patients afflicted worldwide. Fundamental challenges are the complexity of measuring pain appropriately, and the many associated possible confounders. Over the last decades, gender of the investigator has been identified as a conceivable bias in the assessment and management of pain in experimental, as well as, clinical research. However, to the investigators knowledge this issue has not so far been systematically investigated in a postoperative setting.

The objective of this study was to investigate whether the gender of the investigator has an impact on the reported levels of pain intensity after acute or scheduled surgery.

In this prospective paired cross-over study, two investigators of opposite gender independently obtained individually reported pain intensity levels in each study patient based on three different methods of pain assessment the Visual Analogue Scale (VAS), the Numeric Rating Scale (NRS), and the Painmatcher® (PM) technique based on electrical stimulation, in a postoperative study setting at a large urban university hospital in southern Sweden.

DETAILED DESCRIPTION:
Study design This prospective paired clinical cross-over study was carried out in three different Post Anaesthesia Care Units (PACUs) at Skåne University Hospital in Malmö, Sweden. All patients were supervised and managed according to the local standard of care. The measurements were accomplished during daytime over a ten-week study period.

Two investigators, one male and one female, performed the measurements and collected the study data. They were both senior medical students at the same level and of similar age (30 and 38 years, respectively). Postoperative levels of individual pain intensity were obtained as early after arrival at the PACU as possible, depending on how soon the study patient was alert enough to participate. Pain was evaluated in each study patient at two consecutive study sessions at approximately 15-minute intervals, according to a predefined study protocol. Half of the study participants were first evaluated by the female and then by the male investigator, and the other half the other way around, according to a cross-over study design.

Pain evaluation Postoperative pain intensity was assessed with three different study techniques in each study patient.

The Visual Analogue Scale (VAS), is a long-established technique for measuring pain and consists of a 100-millimetre scale ranging from 0 (no pain at all) to 100 (worst imaginable pain). Individual scores were recorded with one decimal number (range 0-10.0).

The Numeric Rating Scale (NRS) is another well-known and reliable method for evaluating pain in clinical practice. The rating is verbal, and the subject is asked to estimate current pain intensity on an 11-point scale, where 0 indicates no pain at all and 10 the worst imaginable pain. The study patients were asked to choose integers only, and no decimal numbers were recorded.

The Painmatcher® (PM) is a rather new instrument (CEFAR Medical AB, Lund, Sweden) developed for assessment of pain with a mild electrical stimulus.

The study patients were told to press two rubber electrodes of the device between their thumb and index finger and to release them as soon as the gradually increasing systaltic sensations in the finger tips induced by electrical current were considered comparable to their current intensity of postoperative pain. On release of the buttons, the local pain immediately ceases and a corresponding integer-based score is displayed on the device. Each patient went through three measurements with the device during each study session.

Study procedures Each study session started with a short interview, where the study participants were asked to shortly describe, in words of their own, the main character of their postoperative pain. They were then requested to rate their current intensity level of pain with the three different study techniques (VAS, PM and NRS in mentioned order). The study patients were equally informed verbally on how to carry out the pain measurements and were blinded to the study aim (of evaluating potential impact of investigator gender). Additional information on surgical and anaesthetic procedures, including current analgesic medication, was obtained from the peri-operative database of the hospital, and from individual patient records.

ELIGIBILITY:
Inclusion Criteria:

* Ongoing PACU care after recent surgery, cognitive and linguistic abilities to understand instructions and participate in the study, and perceived postoperative pain.

Exclusion Criteria:

* Fulfilled inclusion criteria but decline to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2018-09-11 (Actual); Primary Completion 2018-11-16 (Actual); Study Completion 2018-11-16 (Actual)

PRIMARY OUTCOMES:
Postoperative pain assessment with visual analogue scale (VAS). | From arrival at the PACU until approximately 15-minutes after arrival.
  The Visual Analogue Scale (VAS), a 101-point scale for evaluating pain which consists of a 100-millimetre scale ranging from 0 (no pain at all) to 100 (worst imaginable pain). Individual scores were recorded with one decimal number (range 0-10.0).
Postoperative pain assessment with numeric rating scale (NRS). | From arrival at the PACU until approximately 15-minutes after arrival.
  The Numeric Rating Scale (NRS) for evaluating pain. The rating is verbal, and the subject is asked to estimate current pain intensity on an 11-point scale, where 0 indicates no pain at all and 10 the worst imaginable pain.
Postoperative pain assessment with Painmatcher® (PM). | From arrival at the PACU until approximately 15-minutes after arrival.
  The Painmatcher® (CEFAR Medical AB, Lund, Sweden) is an instrument developed for assessment of pain using a mild electrical stimulus, until this pain correlates to the pain already experienced for example postoperative pain.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Sellgren Engskov, PhD student, Principal Investigator — IKVM, Lund University; Jonas Åkeson, Professor, Principal Investigator — IKVM, Lund University
Locations (1):
- Three Post Anaesthesia Care Units (PACUs) at Skåne University Hospital in Malmö, Sweden, Malmo, Sweden

REFERENCES:
- [Derived] Engskov AS, Ydrefors A, El-Jaleb K, Akeson J. Prospective paired crossover evaluation of potential impact of investigator gender on perceived pain intensity early after acute or scheduled surgery. Biol Sex Differ. 2023 Apr 25;14(1):23. doi: 10.1186/s13293-023-00508-9. PMID 37095547

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-01): https://cdn.clinicaltrials.gov/large-docs/97/NCT03968497/Prot_SAP_000.pdf